CLINICAL TRIAL: NCT06001489
Title: The Effects of 360-degree Virtual Reality on Pre-procedural Anxiety in Patients Awaiting Elective Cardiac Surgery Involving a Sternotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Jolanda Kluin, Professor of Cardiothoracic Surgery, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NL2023.22.265
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Cardiac Valve Disease; Aortic Valve Disease; Mitral Valve Disease; Tricuspid Valve Disease
MeSH Terms: conditions — Heart Valve Diseases; Aortic Valve Disease

STUDY DESIGN:
Intervention Model Description: This prospective, single-center, randomized controlled trial (RCT) includes patients awaiting elective open heart surgery via a sternotomy. Patients who met the inclusion criteria were invited to participate in the study. Patients were allocated randomly to either the control or intervention group. The control group received oral information from the treating cardiothoracic surgeon. The intervention group received additional information through an educational 360-degree semi-immersive Virtual Reality (VR) Tour. The VR Tour provided patients a comprehensive visual experience of the entire clinical pathway of the scheduled surgical procedure,
  Patients complete two validated questionnaires immediately following their outpatient clinic visit to assess pre-procedural anxiety. This data was considered the 'baseline'. One day prior to the surgery, during the hospital admission, patients are asked to complete the same questionnaires again. This data will be referred to as 'follow-up (FU)'.
Who Masked: Care Provider
Masking Description: Prior to visiting the outpatient clinic, patients are unaware about their allocation. Only after their outpatient clinic visit, patients are informed about whether they belong to the control or intervention group. The surgeon, nurses OR assistants, however, are not informed about the treatment allocation. This is only known to the investigators and outcomes assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): This patient group received A standard form of patient education, consisting of oral information and an informative flyer during their outpatient clinic visit. After this visit, patients were asked to fill out 2 validated questionnaires: Spielberger's State-Trait Anxiety Inventory (STAI) and the Amsterdam Preoperative Anxiety and Information Scale (APAIS).
  1 day prior to surgery, during admission to the hospital, patients were asked to fill out the STAI and APAIS again.
  Interventions: Diagnostic Test: State Trait Anxiety Inventory; Diagnostic Test: Amsterdam Preoperative Anxiety and Information Scale
- Intervention group - VR (Experimental): This patient group first received a standard form of patient education, consisting of oral information and an informative flyer. Additionally, patients watched a 360-degree VR Tour using a Pico G2 4K VR headset, describing their entire clinical pathway in more detail.
  After this visit, patients were asked to fill out 2 validated questionnaires: Spielberger's State-Trait Anxiety Inventory (STAI) and the Amsterdam Preoperative Anxiety and Information Scale (APAIS).
  1 day prior to surgery, during admission to the hospital, patients were asked to fill out the STAI and APAIS again.
  Interventions: Behavioral: 360-degree Virtual Reality Patient Tour; Diagnostic Test: State Trait Anxiety Inventory; Diagnostic Test: Amsterdam Preoperative Anxiety and Information Scale

INTERVENTIONS:
Behavioral: 360-degree Virtual Reality Patient Tour — A 360-degree video that encompasses the entire clinical pathway. Patients are able to familiarize themselves with the hospital settings (nursery ward, operating room, intensive care unit).
  Arms: Intervention group - VR
Diagnostic Test: State Trait Anxiety Inventory — Spielberger's State Trait Anxiety Inventory provides insight in the presence of anxiety.
  Other Names: STAI
Diagnostic Test: Amsterdam Preoperative Anxiety and Information Scale — This validated questionnaire provides insight in the presence of anxiety. It also measures the need for information.
  Other Names: APAIS

SUMMARY:
Rationale: Patients awaiting cardiac surgery can experience pre-procedural anxiety. This anxiety is associated with increased analgesic needs, increased risk of mortality and prolonged recovery time. Adequate patient education can help diminish pre-procedural anxiety and minimize postoperative complications. Recent studies have demonstrated that Virtual Reality (VR) can function as a useful tool to diminish pre-procedural anxiety in several medical fields. Especially 360 degree VR could familiarize patients with their clinical pathway. Nevertheless, limited to no research on the application of 360 degree VR has been conducted in the context of cardiothoracic surgery yet.

Objective: The aim of this study is to explore the effects and possible benefits of 360 degree VR on pre-procedural anxiety in patients awaiting elective cardiac surgery involving a sternotomy, compared to standard forms of patient education.

Study design: Single-center, randomized controlled trial

Study population: Patients aged 18 or older awaiting elective cardiac surgery involving a sternotomy.

DETAILED DESCRIPTION:
Patients undergoing cardiothoracic surgery are inclined to experience a form of pre-procedural anxiety. Not only can these feelings of concern cause huge psychological discomfort for patients awaiting surgery, but this can also translate into somatic complications, especially for patients with coronary artery disease. These adverse events include a prolonged recovery time, increased risk of re-hospitalization and death amongst other implications and underline the necessity of addressing pre-procedural anxiety. Several approaches have been introduced in an attempt to contain these feelings of concern. Examples that have been applied in the field of surgery include pharmacological interventions as well as extensive patient education. Especially the latter has recently been proven to be effective in diminishing pre-procedural anxiety.

A recent study highlighted the significance of 360-degree Virtual Reality patient education in limiting pre-procedural anxiety levels in patients undergoing percutaneous atrial septal closure. Their research demonstrated that thorough patient education using VR could prevent elevated scores of anxiety, possibly contributing to a diminished number of adverse events in this patient group. Alongside this study, several other researches have hinted at success or are investigating the benefit of VR in managing anxiety levels.

Considering these promising results, the aim of the VR Patient Journey Trial is to evaluate the additional value of 360-degree Virtual Reality as a new modality in reducing pre-procedural anxiety in comparison with regular forms of patient education in patients undergoing coronary artery bypass grafting (CABG) procedures. This procedure remains the most performed type of cardiac surgery and accounts for a large homogenous patient group; an estimated 85% of procedures concern isolated CABG. Managing anxiety levels in this patient group can therefore greatly impact the overall level of patient well-being in cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients awaiting elective cardiac surgery involving a sternotomy
* 18 years or older

Exclusion Criteria:

* Under the age of 18
* History of previous cardiac surgery
* (concomitant) aortic surgery
* Cardiac surgery for congenital heart defects
* Hearing or visual impairments
* Language barriers (inability to understand, speak or read Dutch)
* History of severe mental or psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
State-Anxiety at baseline | During outpatient clinic visit, prior to surgery
  State Anxiety (derived from Spielberger's State-Trait Anxiety Inventory) during outpatient clinic visit prior to surgery. Minimum score value 0, maximum score value 63. Lower outcome means less anxiety, higher outcome means worse anxiety.
Trait-Anxiety at baseline | During outpatient clinic visit, prior to surgery
  Trait Anxiety (derived from Spielberger's State-Trait Anxiety Inventory) during outpatient clinic visit prior to surgery. Minimum score value 0, maximum score value 63. Lower outcome means less anxiety, higher outcome means worse anxiety.
Trait-Anxiety at follow-up | 1 day prior to surgery
  Trait Anxiety (derived from Spielberger's State-Trait Anxiety Inventory) during admission to hospital (1 day prior to surgery). Minimum score value 0, maximum score value 63. Lower outcome means less anxiety, higher outcome means worse anxiety.
State-Anxiety at follow-up | 1 day prior to surgery
  State Anxiety (derived from Spielberger's State-Trait Anxiety Inventory) during admission to hospital (1 day prior to surgery). Minimum score value 0, maximum score value 63. Lower outcome means less anxiety, higher outcome means worse anxiety.
Need-for-information at baseline | During outpatient clinic visit, prior to surgery
  Need for information (derived from Amsterdam Preoperative Anxiety and Information Scale) during outpatient clinic visit prior to surgery. Minimum score value 4, maximum value 20. Lower outcome means less anxiety, higher outcome means worse anxiety.
Need-for-information at follow-up | 1 day prior to surgery
  Need for information (derived from Amsterdam Preoperative Anxiety and Information Scale) during outpatient clinic visit prior to surgery. Minimum score value 4, maximum value 20. Lower outcome means less anxiety, higher outcome means worse anxiety.
Pre-procedural anxiety at baseline | During outpatient clinic visit, prior to surgery
  Pre-procedural anxiety (derived from Amsterdam Preoperative Anxiety and Information Scale) during outpatient clinic visit prior to surgery. Minimum score value 4, maximum value 20. Lower outcome means less anxiety, higher outcome means worse anxiety.
Pre-procedural anxiety at follow-up | 1 day prior to surgery
  Pre-procedural anxiety (derived from Amsterdam Preoperative Anxiety and Information Scale) during outpatient clinic visit prior to surgery. Minimum score value 4, maximum value 20. Lower outcome means less anxiety, higher outcome means worse anxiety.
HR at baseline | During outpatient clinic visit, prior to surgery
  Heartrate in bpm (beats per minute) during outpatient clinic visit prior to surgery
HR at follow-up | 1 day prior to surgery
  Heartrate in bpm (beats per minute) during admission to hospital (1 day prior to surgery)
HR in operation room | in the OR on the day of surgery
  Heartrate in bpm (beats per minute) in the operation room on the day of surgery
Diastolic blood pressure at baseline | During outpatient clinic visit prior to surgery
  Diastolic blood pressure (in mm/Hg) during outpatient clinic visit prior to surgery
Systolic blood pressure at baseline | During outpatient clinic visit prior to surgery
  Systolic blood pressure (in mm/Hg) during outpatient clinic visit prior to surgery
Diastolic blood pressure at follow-up | 1 day prior to surgery
  Diastolic blood pressure (in mm/Hg) during admission to hospital (1 day prior to surgery)
Systolic blood pressure at follow-up | 1 day prior to surgery
  Systolic blood pressure (in mm/Hg) during admission to hospital (1 day prior to surgery)
Diastolic blood pressure in OR | in the OR on the day of surgery
  Systolic blood pressure (in mm/Hg) in the operation room on the day of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jolanda Kluin, MD, PhD, Principal Investigator — j.kluin@amsterdamumc.nl
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
When asked for, a construction will be made to share data. At the end of the study.